CLINICAL TRIAL: NCT06937918
Title: Effect of Dynamic Arterial Elastance and Assisted Fluid Management Software Guided Adjustment of Vasopressor and Fluid Therapy in Septic Shock Resuscitation; A Pilot Study
Brief Title: Effect of Dynamic Arterial Elastance and Assisted Fluid Management Software Guided Resuscitation in Septic Shock: Pilot Study
Acronym: DAFM shock
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SI 118/2025
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Critical Illness; Fluid Over-load; Dynamic Arterial Elastance; Septic Shock
Keywords: critical illness; dynamic arterial elastance; stroke volume change prediction; fluid overload; ischemic complication; septic shock
MeSH Terms: conditions — Critical Illness; Shock, Septic; Edema

STUDY DESIGN:
Intervention Model Description: A fluid challenge using a stroke volume change prediction (∆SVpredict) and Eadyn guide. If the ∆SVpredict is more than 10%, isotonic crystalloid of 500 ml will be administered in 30 minutes, and wait for the response of the machine for 5 minutes after loading. If ∆SVpredict is still more than 10%, continuous fluid loading was reapplied until SVV was less than 10% (fluid therapy will be stopped if ∆SVpredict is less than 10%) and dynamic arterial elastance (EAdyn) reaches the goal of 0.8-1.0[5] along with a vasopressor will be administered and titrated every 10 minutes until the target mABP > 65 mmHg is reached.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the standard of care group (Active Comparator): The standard of care group will be treated according to according to septic shock guidelines 2021; In brief A vasopressor with optimal ideal fluid (at least 30 ml/kg) will be given to achieve the hemodynamic target (MAP ≥ 65 mm Hg) by fluid challenge technique guided by MAP and central venous pressure (CVP) changes after fluid challenge. Fluid-responsive tests can be used as a subsidiary, depending on the attending physician. Early Norepinephrine (NE) infusion can be used with a standard dose of 0.05 mcg/k/min and titrated at the rate of 0.01-0.02 mcg/kg/min every 10 min until 0.25 mcg/kg/min was achieved; then, the second line vasopressor will be added and adjusted to the target of vasopressor. Hydrocortisone can be given according to septic shock guidelines.
  Interventions: Other: The standard care for septic shock
- AFM and Eadyn - guided resuscitation group (Experimental): Patients randomized to this arm are treated with the standard of care for patients with septic shock as described for 'the standard of care' arm, along with the AFM and Eadyn - guided resuscitation group, as detailed under 'Interventions'
  Interventions: Device: The AFM and Eadyn - guided resuscitation group; Other: The standard care for septic shock

INTERVENTIONS:
Device: The AFM and Eadyn - guided resuscitation group — A fluid challenge using a stroke volume change prediction (∆SVpredict) and Eadyn guide. If the ∆SVpredict is more than 10%, isotonic crystalloid of 500 ml will be administered in 30 minutes, and the machine's response will be awaited. If ∆SVpredict is still more than 10%, continuous fluid loading was reapplied until SVV was less than 10% (fluid therapy will be stopped if ∆SVpredict is less than 10%) and dynamic arterial elastance (EAdyn) reaches the goal of 0.8-1.0 along with a vasopressor will be administered and titrated every 10 minutes until the target MAP > 65 mmHg is reached. After MAP of 65 achieved, tissue perfusion including urine output, capillary refill time, and serum lactate will be assessed
  Other Names: hemosphere; dynamic arterial elastance
  Arms: AFM and Eadyn - guided resuscitation group
Other: The standard care for septic shock — The standard of care group will be treated according to according to septic shock guidelines 2021; In brief A vasopressor with optimal ideal fluid (at least 30 ml/kg) will be given to achieve the hemodynamic target (MAP ≥ 65 mm Hg) by fluid challenge technique guided by MAP and central venous pressure (CVP) changes after fluid challenge. Fluid-responsive tests can be used as a subsidiary, depending on the attending physician. Early Norepinephrine (NE) infusion can be used with a standard dose of 0.05 mcg/k/min and titrated at the rate of 0.01-0.02 mcg/kg/min every 10 min until 0.25 mcg/kg/min was achieved; then, the second line vasopressor will be added and adjusted to the target of vasopressor. Hydrocortisone can be given according to septic shock guidelines.
  After MAP of 65 achieved, tissue perfusion including urine output, capillary refill time, and serum lactate will be assessed

SUMMARY:
To investigate the benefit of using the AFM and Eadyn-guided fluid and vasopressor therapy in septic shock resuscitation for mechanically ventilated patients compared with the standard of care. The investigators hypothesize that using the AFM and Eadyn-guided fluid/vasopressor titration in septic shock patients who underwent mechanical ventilation might reduce the time to shock reversal.

DETAILED DESCRIPTION:
Hypotension in the context of an intensive care unit has been associated with a higher risk of death and multiorgan dysfunction. Vascular leakage and systemic vasodilatation are brought on by systemic inflammation from infections. These are the hallmarks of septic shock in which 90% of cases of shock are mostly distributive and hypovolemic. Early vasopressors and fluid therapy are increasingly used at the start of vasodilatory shock resuscitation since this method improves the rate of shock control within 6 hours in septic shock resuscitation. Norepinephrine is the first-line vasopressor for vasodilatory shock. However, resuscitation with an accurate amount of fluid and vasopressor is challenging in clinical practice. Fluid overload and overuse of vasopressors are prevalent and increase mortality. Together with a higher dose of norepinephrine, it may increase the risk of ischemic complications.

A new hemodynamic monitoring device (Hemosphere(R) - Edward Lifescience, California, USA) provides two novel parameters for hemodynamic monitoring: the new device with artificial intelligence developed by a retrospective cohort (used for training) and a prospective (local hospital cohort used for external validation). The feature of Hemosphere(R), including dynamic arterial elastance (Eadyn) and stroke volume change prediction (∆SVpredict) as the assist fluid management (AFM) based on arterial pressure waveform analysis by the monitoring software, was detected in arterial line waveform without any complication of a safety issue.

The ratio of pulse pressure to stroke volume (PP/SV) is defined by dynamic arterial elastance (Eadyn), the reciprocal of compliance within the range of 0.8 to 1.0 is the optimization of arterial load that can predict arterial pressure response to fluid administration and vasopressor weaning. The prediction of the stroke volume changes following the upcoming fluid therapy (∆SVpredict) uses stroke volume variation parameters and closed-loop feedback data, which should be less than 10% to indicate optimal fluid administration. Consequently, this technique offers a useful means of evaluating arterial tone related to preload responsiveness parameters predicting the hemodynamic response to increases in cardiac preload.

However, several studies show the benefit of this tool in perioperative patients, and the evidence on the benefit of using this monitoring to guide septic shock resuscitation is limited. In a previous study, Eadyn can predict a decrease in mean arterial pressure linked to a reduction in norepinephrine dosage. This study aimed to investigate the benefit of using AFM and Eadyn-guided fluid and vasopressor therapy in septic shock resuscitation compared with the standard of care

ELIGIBILITY:
Inclusion Criteria:

* All Thai consecutive patients older than 18 years with a diagnosis of sepsis or septic shock in medical ICU, defined by clinically suspected or confirmed infection and MAP <65 mmHg according to the criteria of the Surviving Sepsis Campaign 2021(11)with onset of shock in less than 24 hours.
* Already receiving or planning for mechanical ventilation
* Already receiving or planning for arterial catheter placement for invasive arterial pressure monitoring
* All patients will receive an echocardiogram with a cut point of LVEF > 30% to be included in the study

Exclusion Criteria:

* Active, immediate, life-threatening cardiac arrhythmia, defined as ventricular tachycardia and ventricular fibrillation
* Acute cerebral vascular event, including both acute ischemic stroke or intracranial hemorrhage
* Acute coronary syndrome
* cardiogenic shock, acute heart failure
* Severe asthma exacerbation
* Fluid intolerance: hypoxemia (P:F ratio < 150)
* Life-threatening gastrointestinal hemorrhage
* Pregnancy
* Requirement for immediate surgery within 2 hours of randomization
* Advanced-stage cancer with predicted survival of less than 6 months
* Oliguric AKI with signs of volume overload

Withdrawal or termination criteria

* The patient and legal representative request for withdrawal
* The attending physician requested a withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-23 (Estimated); Primary Completion 2027-04-08 (Estimated); Study Completion 2028-04-08 (Estimated)

PRIMARY OUTCOMES:
time to shock reversal | 28 days
  the time from diagnosis of septic shock until the achievement of sustained MAP of ≥65 mmHg with evidence of adequate tissue perfusion (continuation of urine ﬂow ≥ 0.5 ml/kg/h or normalized or continuing decrease in serum lactate ≥10% from the previous value) without any vasopressor infusion

SECONDARY OUTCOMES:
a time-to-goal achievement for septic shock resuscitation | 28 days
  MAP ≥ 65 mmHg with vasopressors and optimized tissue perfusion
time to NE titrating | 48 hours
maximum dose of vasopressors | 48 hours
volume of fluid therapy during resuscitation | 48 hours
fluid before randomization | 48 hours
fluid accumulation at 24 hours | 24 hours
fluid accumulation at 72 hours | 72 hours
fluid accumulation at 7 days | 7 days
28-day hospital mortality | 28 days
ICU length of stay | 28 days
hospital length of stay | 28 days
shock reversal at 6 hours | 6 hours
  Shock reversal is defined as mean arterial pressure at or more than 65 mmHg with one of the following: -Reduction of serum lactate level of 20% or more -Hourly urine output of 0.5 mL/kg or more
rate of new initiation of renal replacement therapy | 28 days
time to initiation of renal replacement therapy | 28 days
Vasopressor-free day | 28 days
  Number of days that patient is alive after successful discontinuation of vasoactive agents in the first 28 days, with the day of randomization defined as Day 1. Successful discontinuation of vasoactive agents is defined as discontinuation of vasoactive agents without resumption until Day 28 or until hospital discharge, whichever is first. In case of multiple periods of vasoactive agents use, the days from the final discontinuation of vasoactive agents are counted. All 28-day non-survivors are counted as 0, irrespective of their use of vasoactive agents at the time of death, and censored observations after 28 days
Ventilator-free day | 28 days
  Number of days that patient is alive after successful liberation of mechanical ventilation in the first 28 days, with the day of randomization defined as Day 1. Successful liberation of mechanical ventilation is defined as the discontinuation of mechanical ventilation (either via orotracheal or tracheostomy tube) for 48 hours or more. Non-invasive positive pressure ventilation is not regarded as mechanical ventilation. In case of multiple periods of mechanical ventilation, the days from the final successful liberation of mechanical ventilation within 28 days are counted. All 28-day non-survivors are counted as 0, irrespective of their ventilation status at the time of death, and censored observations after 28 days
Renal replacement therapy(RRT)-free day | 28 days
  Number of days that patient is alive after successful discontinuation of renal-replacement therapy in the first 28 days, with the day of randomization defined as Day 1. Successful discontinuation of renal-replacement therapy is defined as discontinuation of all modes of renal-replacement therapy without resumption for at least 7 days and until Day 28 or until hospital discharge, whichever is first. Hemoperfusion according to treatment protocol in 'Standard of care and hemoperfusion with HA-330' arm is not counted as renal-replacement therapy. All 28-day non-survivors are counted as 0, irrespective of their use of renal-replacement therapy at the time of death, and censored observations after 28 days
Serum lactate at 0 hours, 1 hour, and 6 hours | 6 hours

OTHER OUTCOMES:
adverse event | 28 days
  ischemic complication and arrhythmia

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital, Bangkok Noi, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asfar P, Meziani F, Hamel JF, Grelon F, Megarbane B, Anguel N, Mira JP, Dequin PF, Gergaud S, Weiss N, Legay F, Le Tulzo Y, Conrad M, Robert R, Gonzalez F, Guitton C, Tamion F, Tonnelier JM, Guezennec P, Van Der Linden T, Vieillard-Baron A, Mariotte E, Pradel G, Lesieur O, Ricard JD, Herve F, du Cheyron D, Guerin C, Mercat A, Teboul JL, Radermacher P; SEPSISPAM Investigators. High versus low blood-pressure target in patients with septic shock. N Engl J Med. 2014 Apr 24;370(17):1583-93. doi: 10.1056/NEJMoa1312173. Epub 2014 Mar 18. PMID 24635770
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Hylander Moller M, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. Crit Care Med. 2021 Nov 1;49(11):e1063-e1143. doi: 10.1097/CCM.0000000000005337. No abstract available. PMID 34605781
- [Background] Maheshwari K, Malhotra G, Bao X, Lahsaei P, Hand WR, Fleming NW, Ramsingh D, Treggiari MM, Sessler DI, Miller TE; Assisted Fluid Management Study Team. Assisted Fluid Management Software Guidance for Intraoperative Fluid Administration. Anesthesiology. 2021 Aug 1;135(2):273-283. doi: 10.1097/ALN.0000000000003790. PMID 33901281
- [Background] Kelly RP, Ting CT, Yang TM, Liu CP, Maughan WL, Chang MS, Kass DA. Effective arterial elastance as index of arterial vascular load in humans. Circulation. 1992 Aug;86(2):513-21. doi: 10.1161/01.cir.86.2.513. PMID 1638719
- [Background] Lai CJ, Cheng YJ, Han YY, Hsiao PN, Lin PL, Chiu CT, Lee JM, Tien YW, Chien KL. Hypotension prediction index for prevention of intraoperative hypotension in patients undergoing general anesthesia: a randomized controlled trial. Perioper Med (Lond). 2024 Jun 15;13(1):57. doi: 10.1186/s13741-024-00414-7. PMID 38879506
- [Background] Dong S, Wang Q, Wang S, Zhou C, Wang H. Hypotension prediction index for the prevention of hypotension during surgery and critical care: A narrative review. Comput Biol Med. 2024 Mar;170:107995. doi: 10.1016/j.compbiomed.2024.107995. Epub 2024 Jan 18. PMID 38325215
- [Background] Guinot PG, Bernard E, Levrard M, Dupont H, Lorne E. Dynamic arterial elastance predicts mean arterial pressure decrease associated with decreasing norepinephrine dosage in septic shock. Crit Care. 2015 Jan 19;19(1):14. doi: 10.1186/s13054-014-0732-5. PMID 25598221
- [Background] Monge Garcia MI, Jian Z, Settels JJ, Hunley C, Cecconi M, Hatib F, Pinsky MR. Performance comparison of ventricular and arterial dP/dtmax for assessing left ventricular systolic function during different experimental loading and contractile conditions. Crit Care. 2018 Nov 29;22(1):325. doi: 10.1186/s13054-018-2260-1. PMID 30486866
- [Background] Zhou X, Pan W, Chen B, Xu Z, Pan J. Predictive performance of dynamic arterial elastance for arterial pressure response to fluid expansion in mechanically ventilated hypotensive adults: a systematic review and meta-analysis of observational studies. Ann Intensive Care. 2021 Jul 31;11(1):119. doi: 10.1186/s13613-021-00909-2. PMID 34331607
- [Background] Kouz K, Monge Garcia MI, Cerutti E, Lisanti I, Draisci G, Frassanito L, Sander M, Ali Akbari A, Frey UH, Grundmann CD, Davies SJ, Donati A, Ripolles-Melchor J, Garcia-Lopez D, Vojnar B, Gayat E, Noll E, Bramlage P, Saugel B. Intraoperative hypotension when using hypotension prediction index software during major noncardiac surgery: a European multicentre prospective observational registry (EU HYPROTECT). BJA Open. 2023 May 4;6:100140. doi: 10.1016/j.bjao.2023.100140. eCollection 2023 Jun. PMID 37588176
- [Background] Monge Garcia MI, Gil Cano A, Gracia Romero M. Dynamic arterial elastance to predict arterial pressure response to volume loading in preload-dependent patients. Crit Care. 2011;15(1):R15. doi: 10.1186/cc9420. Epub 2011 Jan 12. PMID 21226909
- [Background] Hatib F, Jian Z, Buddi S, Lee C, Settels J, Sibert K, Rinehart J, Cannesson M. Machine-learning Algorithm to Predict Hypotension Based on High-fidelity Arterial Pressure Waveform Analysis. Anesthesiology. 2018 Oct;129(4):663-674. doi: 10.1097/ALN.0000000000002300. PMID 29894315
- [Background] Messmer AS, Zingg C, Muller M, Gerber JL, Schefold JC, Pfortmueller CA. Fluid Overload and Mortality in Adult Critical Care Patients-A Systematic Review and Meta-Analysis of Observational Studies. Crit Care Med. 2020 Dec;48(12):1862-1870. doi: 10.1097/CCM.0000000000004617. PMID 33009098
- [Background] Permpikul C, Tongyoo S, Viarasilpa T, Trainarongsakul T, Chakorn T, Udompanturak S. Early Use of Norepinephrine in Septic Shock Resuscitation (CENSER). A Randomized Trial. Am J Respir Crit Care Med. 2019 May 1;199(9):1097-1105. doi: 10.1164/rccm.201806-1034OC. PMID 30704260
- [Background] Angus DC, van der Poll T. Severe sepsis and septic shock. N Engl J Med. 2013 Aug 29;369(9):840-51. doi: 10.1056/NEJMra1208623. No abstract available. PMID 23984731
- See also: sample size — https://doi.org/10.48550/arXiv.2105.05483